CLINICAL TRIAL: NCT01582672
Title: An International Phase 3 Randomized Trial of Autologous Dendritic Cell Immunotherapy (AGS-003) Plus Standard Treatment of Advanced Renal Cell Carcinoma (ADAPT)
Brief Title: Phase 3 Trial of Autologous Dendritic Cell Immunotherapy Plus Standard Treatment of Advanced Renal Cell Carcinoma
Acronym: ADAPT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Argos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGS-003-007; 2012-000871-17 (EudraCT Number)
Record Dates: First submitted 2012-04-19; First posted 2012-04-23 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2017-06

CONDITIONS: Advanced Renal Cell Carcinoma; Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma
Keywords: RCC; Kidney Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AGS-003 + Standard Treatment (Experimental): Subjects on this arm will receive standard treatment for Renal Cell Carcinoma. In addition, subjects will receive AGS-003.
  Interventions: Biological: AGS-003
- Standard Treatment (Active Comparator): Subjects on this arm will receive standard treatment for Renal Cell Carcinoma.
  Interventions: Drug: Standard Treatment

INTERVENTIONS:
Drug: Standard Treatment — Standard treatment for Renal Cell Carcinoma
  Other Names: Sunitinib
  Arms: Standard Treatment
Biological: AGS-003 — Autologous Dendritic Cell product. Intradermal injections; 8 injections in the 1st year followed by quarterly boosters.
  Arms: AGS-003 + Standard Treatment

SUMMARY:
This is a trial of AGS-003, which is being studied as a possible treatment for Advanced Renal Cell Carcinoma. The purpose of this study is to determine whether there is an overall survival (OS) benefit between subjects treated with AGS-003 in combination with standard treatment versus subjects treated with standard treatment alone.

DETAILED DESCRIPTION:
This study will investigate the combination of an autologous ribonucleic acid (RNA) electroporated dendritic cell (DC) based immunotherapy, AGS-003, plus standard treatment (initiating with sunitinib). The primary objective in this study is to determine the median OS achieved by this combination compared to the OS resulting from use of active control (standard treatment), in a population of adults with advanced renal cell carcinoma (RCC), with nephrectomy indicated, and with remaining metastatic disease.

ELIGIBILITY:
Key Inclusion Criteria for Tumor Collection:

1. Diagnosis or clinical signs of advanced RCC
2. Scheduled for cytoreductive or partial nephrectomy

Key Exclusion Criteria for Tumor Collection:

1. Known inability to undergo sunitinib treatment as currently labeled, due to pre-existing medical conditions
2. Requirement for systemic chronic immunosuppressive drugs or corticosteroids
3. Evidence of brain metastases prior to nephrectomy

Key Inclusion Criteria for Treatment Study:

1. Advanced disease, histologically assessed as RCC, with predominantly clear cell histology
2. Metastatic disease (measurable or non-measurable) that can be monitored throughout the course of the study participation per RECIST 1.1
3. Subjects who are candidates for standard first-line therapy initiating with sunitinib
4. Time from diagnosis to treatment < 1 year
5. Karnofsky performance status (KPS) ≥ 70%
6. Life expectancy of 6 months or greater
7. Resolution of all acute toxic effects of prior radiotherapy or surgical procedures to Grade ≤ 1 according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
8. Adequate hematologic, renal, hepatic, and coagulation function
9. Negative serum pregnancy test for female subjects with reproductive potential, and agreement of all male and female subjects of reproductive potential to use a reliable form of contraception during the study and for 12 weeks after the last dose of study drug
10. Normal ECG or clinically non-significant finding(s) at Screening
11. Able to abstain from taking prohibited drugs, either prescription or non-prescription, during the treatment phase of the study
12. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Key Exclusion Criteria for Treatment Study:

1. Prior systemic therapy (including adjuvant or neoadjuvant) of any kind for RCC, including immunotherapy, chemotherapy, hormonal, or investigational therapy
2. Prior history of malignancy within the preceding 3 years, except for adequately treated in situ carcinomas or non-melanoma skin cancer, adequately treated early stage breast cancer, superficial bladder cancer, and non-metastatic prostate cancer with a normal PSA
3. History of or known brain metastases, spinal cord compression, or carcinomatous meningitis, or evidence of brain or leptomeningeal disease
4. Patients with 4 or more of the following risk factors:

   1. Hgb < LLN
   2. Corrected calcium > 10.0 mg/dL
   3. KPS < 80%
   4. Neutrophils > ULN
   5. Platelets > ULN
5. Planned or elective surgical treatment post-nephrectomy for the direct management of RCC, within 28 days before Visit 1 (Week 0)
6. NCI CTCAE Grade 3 hemorrhage < 28 days before Visit 1 (Day 0)
7. Clinically significant cardiovascular conditions within 3 months prior to Randomization
8. Significant gastrointestinal abnormalities
9. Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
10. Active autoimmune disease or condition requiring chronic immunosuppressive therapy
11. Clinically significant infections, including human immunodeficiency virus, syphilis, and active hepatitis B or C
12. Current treatment with an investigational therapy on another clinical trial
13. Pregnancy or breastfeeding
14. Any serious medical condition or illness considered by the investigator to constitute an unwarranted high risk for investigational treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2012-11; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From date of subject randomization to date of death; assessed up to 42 months or until 290 deaths have been accrued on study
  Duration from randomization to death

SECONDARY OUTCOMES:
Progression Free Survival | From date of subject randomization to date of progression; assessed up to 42 months
Tumor Response | From date of subject randomization to date of progression; assessed up to 42 months
  Monitor for evidence of the following tumor responses: Objective response rate, Duration of overall response, and Disease control rate.
Monitor treatment emergent adverse events between both arms | From safety baseline until either meeting a discontinuation criterion or death; assessed up to 42 months
  Compare adverse events between both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Figlin, MD, FACP, Principal Investigator — Cedars-Sinai Medical Center; Christopher G Wood, MD, FACP, Principal Investigator — M.D. Anderson Cancer Center
Locations (105):
- United States (74):
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - La Jolla, California
  - Los Angeles, California
  - San Francisco, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Marietta, Georgia
  - Boise, Idaho
  - Meridian, Idaho
  - Chicago, Illinois
  - Maywood, Illinois
  - Springfield, Illinois
  - Greenwood, Indiana
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Wichita, Kansas
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Lansing, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Hackensack, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - East Syracuse, New York
  - New Hyde Park, New York
  - New York, New York
  - Stony Brook, New York
  - Syracuse, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Middletown, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Springfield, Oregon
  - Allentown, Pennsylvania
  - Danville, Pennsylvania
  - Easton, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Myrtle Beach, South Carolina
  - Sioux Falls, South Dakota
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Virginia Beach, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Canada (8):
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - London, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Québec
- Czechia (4):
  - Hradec Králové
  - Liberec
  - Olomouc
  - Prague
- Hungary (2):
  - Budapest
  - Debrecen
- Israel (6):
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Rehovot
  - Tel Litwinsky
  - Ẕerifin
- Italy (2):
  - Roma
  - Rome
- Spain (6):
  - Badalona
  - Barcelona
  - Madrid
  - Seville
  - Valencia
  - Vigo
- United Kingdom (3):
  - Cambridge
  - Norwich
  - Preston

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Figlin RA, Tannir NM, Uzzo RG, Tykodi SS, Chen DYT, Master V, Kapoor A, Vaena D, Lowrance W, Bratslavsky G, DeBenedette M, Gamble A, Plachco A, Norris MS, Horvatinovich J, Tcherepanova IY, Nicolette CA, Wood CG; ADAPT study group. Results of the ADAPT Phase 3 Study of Rocapuldencel-T in Combination with Sunitinib as First-Line Therapy in Patients with Metastatic Renal Cell Carcinoma. Clin Cancer Res. 2020 May 15;26(10):2327-2336. doi: 10.1158/1078-0432.CCR-19-2427. Epub 2020 Feb 7. PMID 32034074